CLINICAL TRIAL: NCT01064778
Title: The Effects of Dietary Glycemic Index on Brain Function
Brief Title: Glycemic Index and Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Children's Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Alsop, Director of MRI Research, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-003
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: Glycemic Index; Brain; Intake Regulation; Weight Loss; Hunger; Diet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low GI (Active Comparator)
  Interventions: Other: Low GI
- High GI (Experimental)
  Interventions: Other: High GI

INTERVENTIONS:
Other: Low GI — Subjects will be instructed to consume a liquid test meal with a low GI over 5 minutes after baseline laboratory evaluations. The low and high GI meal contain similar amounts of milk, oil, dried egg whites, equal, and vanilla extract. The low GI meal corn-starch as a carbohydrate. Both meals have similar macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. The high vs. low GI meals have a predicted difference in GI of 90 vs. 40, and consistent with this prediction, a pilot study in obese young adults found a 2.2-fold difference in glycemic response (p<0.001). The test meals will provide 25% of individual daily energy requirements.
  Arms: Low GI
Other: High GI — Subjects will be instructed to consume a liquid test meal with a high GI over 5 minutes after baseline laboratory evaluations. The low and high GI meal contain similar amounts of milk, oil, dried egg whites, equal, and vanilla extract. The high GI meal contains corn-syrup as a carbohydrate. Both meals have similar macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. The high vs. low GI meals have a predicted difference in GI of 90 vs. 40, and consistent with this prediction, a pilot study in obese young adults found a 2.2-fold difference in glycemic response (p<0.001). The test meals will provide 25% of individual daily energy requirements.
  Arms: High GI

SUMMARY:
The investigators propose examine the effects of the dietary factor glycemic index (GI) on brain areas that control food intake and hunger. This knowledge could help design dietary approaches that decrease hunger, and thus promote new weight loss strategies.

DETAILED DESCRIPTION:
Most individuals have great difficulty following reduced calorie diets because they experience increased hunger. This process is regulated by specific brain areas. Though many psychological and environmental factors are involved, physiological effects of diet may have a significant impact. The postprandial rise in blood glucose, quantified by the glycemic index (GI), is of particular interest. High GI meals elicit hormonal events that limit availability of metabolic fuels, causing hunger and overeating, especially in people with high insulin secretion.

Our aim is to examine how postprandial changes after high versus low GI meals affect hunger and brain function in areas of intake control. Specifically, we speculate that obese individuals will demonstrate functional changes in brain areas of intake control and increased hunger after a high versus low GI meal.

We will recruit obese, young adults and quantify their insulin secretion during a 2-hour oral glucose tolerance test. A brief practice MRI session will serve to familiarize the subjects with the scanning process. During the two test sessions, standardized test meals with high versus low GI will be given in a randomized, blinded cross-over design. Serial blood levels of hormones, metabolic fuels, and metabolites will be correlated with perceived hunger, and a perfusion MRI scan will be performed to assess brain activation during the late postprandial phase, at the nadir of blood sugar and insulin levels (4 hours postprandial).

This work will inform an integrated physiological model relating peripheral postprandial changes to brain function and hunger. In addition, findings may provide evidence of a novel diet-phenotype, in which baseline clinical characteristics can be used to predict which weight loss diet will work best for a specific individual. Metabolite profiling might shed light on the mechanisms linking diet composition to brain function, and provide feasible clinical markers of the identified phenotype to facilitate translation into practice.

ELIGIBILITY:
Inclusion criteria

1. Males age 18 to 35 years
2. BMI less than or equal to 25 for age and gender

Exclusion criteria

1. weight > 300 lbs
2. largest body circumference > 144cm
3. body shape incompatible with MRI scanner or equipment
4. MRI exclusion criteria
5. large fluctuations in body weight (5% over preceding 6 months, 2.5% during the study)
6. known medical problems that may affect metabolism or hormones
7. diabetes mellitus (fasting plasma glucose ≥126 mg/dL)
8. other abnormal laboratory screening tests
9. taking any medications or dietary supplements that might affect body weight, appetite, or energy expenditure
10. smoking or illicit substance abuse
11. high levels of physical activity (>30 minutes per day, > 4days per week)
12. currently following a weight loss diet
13. allergies or intolerance to eggs, vanilla extract, equal, canola oil, milk, cornstarch, corn syrup

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Blood Flow in Brain Areas of Intake Control. | 4 hours postprandial

SECONDARY OUTCOMES:
Subjective Hunger Rating | Every 30 minutes for 5 hours.
Blood Glucose Level | Every 30 minutes for 5 hours.
Blood Insulin Level | Every 30 minutes for 5 hours
Blood Glucagon Level | Every 30 minutes for 5 hours.
Blood Growth Hormone Level | Every 30 minutes for 5 hours.
Blood Epinephrine Level | Every 30 minutes for 5 hours.
Blood Fatty Acids Level | Every 30 minutes for 5 hours.
  measuring metabolite profiles

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; David Alsop, PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Belinda S Lennerz, MD, PhD, Study Director — Boston Children's Hospital
Locations (3):
- United States (3):
  - Children's Hospital Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Lennerz BS, Alsop DC, Holsen LM, Stern E, Rojas R, Ebbeling CB, Goldstein JM, Ludwig DS. Effects of dietary glycemic index on brain regions related to reward and craving in men. Am J Clin Nutr. 2013 Sep;98(3):641-7. doi: 10.3945/ajcn.113.064113. Epub 2013 Jun 26. PMID 23803881